CLINICAL TRIAL: NCT01961882
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase 2 Trial to Evaluate the Efficacy and Safety of OCV-501 in Elderly Patients With Acute Myeloid Leukemia
Brief Title: A Phase 2 Trial to Evaluate the Efficacy and Safety of OCV-501 in Elderly Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Collaborators: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 311-12-001; JapicCTI-142429 (Other: Japan Pharmaceutical Information Center)
Record Dates: First submitted 2013-10-10; First posted 2013-10-14 (Estimated); Results first posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: OCV-501; Acute Myeloid Leukemia; Antigen specific cancer immunotherapeutic
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- OCV-501 arm (Experimental)
  Interventions: Drug: OCV-501
- Placebo arm (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OCV-501
  Arms: OCV-501 arm
Drug: Placebo
  Arms: Placebo arm

SUMMARY:
To compare disease-free survival in patients 60 years or older with acute myeloid leukemia (AML) who are randomly assigned to receive either OCV-501 monotherapy or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML who achieved first complete remission within one or two courses of standard induction therapy, and completed standard consolidation therapy (more than one course).
* Patients who are 60 years or older.
* Patients who have provided written informed consent within 90 days from the last dose of consolidation therapy on an informed consent form that has been approved by an institutional review board or independent ethics committee.

Exclusion Criteria:

* Patients who have acute promyelocytic leukemia (APL) with t(15;17) (q22;q12), (PML/RARA) karyotype abnormalities, and other variant types.
* Patients who are scheduled for hematopoietic stem cell transplantation.
* Patients who have received drugs potentially affecting the immune system within 4 weeks before starting IMP administration or who may receive such drugs after start of the trial.
* Patients who have a severe concurrent disease or psychiatric illness likely to interfere with participation in this trial.
* Patients who are HIV antibody positive, HBV-DNA positive or have unrecovered chronic hepatitis C with positive HCV antibody.
* Patients who have cirrhosis.
* Patients judged to be ineligible by the investigator (or subinvestigator) for any other reasons.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2013-10; Primary Completion 2017-11-16 (Actual); Study Completion 2017-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jun-ichi Hashimoto, PhD, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (14):
- Japan (8):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Shikoku Region
  - Tohoku Region
- South Korea (2):
  - Daegu
  - Seoul
- Taiwan (4):
  - Kaoshiung
  - Taichung
  - Tainan
  - Taipei

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 134 subjects randomized in this trial, one subject who was randomized but did not receive the investigational medicinal product (IMP) was excluded from all analysis data sets.
Groups:
- OCV-501: 3 mg of OCV-501 (0.4 mL) was administered subcutaneously, once-weekly up to the 8th administration, and once every 2 weeks from the 9th administration onward.
- Placebo: Placebo (0.4 mL) was administered subcutaneously, once-weekly up to the 8th administration, and once every 2 weeks from the 9th administration onward.
Period: Overall Study
Arm/Group | OCV-501 | Placebo
Started | 69 | 65
Completed | 19 | 23
Not Completed | 50 | 42
Not completed — Adverse Event | 3 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Relapse of AML | 39 | 37
Not completed — Use of prohibited concomitant drug or therapy | 2 | 2
Not completed — Subject found to be ineligible for the trial after registration | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): all subjects who received the IMP at least once and from whom data on at least 1 efficacy endpoint were obtained after the start of IMP administration.
Groups:
- Total: Total of all reporting groups
Arm/Group | OCV-501 | Placebo | Total
Number analyzed (Participants) | 68 | 65 | 133
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 18 | 37
  >=65 years | 49 | 47 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (5.61) | 68.6 (6.20) | 68.4 (5.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 30 | 52
  Male | 46 | 35 | 81
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 68 | 65 | 133
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 9 | 9 | 18
  Japan | 52 | 53 | 105
  Taiwan | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Disease-Free Survival
Description: Disease-free survival (DFS) was defined as the time from randomization until relapse or death from any cause, whichever came first, by the DFS-cutoff date.
Time Frame: 2 years (treatment period)
Population: FAS: all subjects who received the IMP at least once and from whom data on at least 1 efficacy endpoint were obtained after the start of IMP administration.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OCV-501 | Placebo
Number analyzed (Participants) | 68 | 65
percentage of participants | 40.9 [28.2 to 53.2] | 41.4 [28.9 to 53.5]

2. Secondary Outcome: Overall Survival
Description: Subjects were surveyed for survival by the date of cutoff. The cutoff date was set as the date after 728 days (2 years) from the day that the last subject started IMP administration.
Time Frame: 2 years (treatment period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OCV-501 | Placebo
Number analyzed (Participants) | 68 | 65
percentage of participants | 60.3 [47.7 to 70.8] | 58.5 [45.6 to 69.3]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from the first dose of IMP to post-treatment observation (up to 17 days after the last dose of IMP or within 7 days from withdrawal judgment).
Arm/Group | OCV-501 | Placebo
All-Cause Mortality (participants affected / at risk) | 1/68 | 1/65
Serious Adverse Events (participants affected / at risk) | 7/68 | 7/65
Other Adverse Events (participants affected / at risk) | 67/68 | 59/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OCV-501 (N=68) | Placebo (N=65)
Infectious colitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypoglycaemic encephalopathy (Nervous system disorders) | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OCV-501 (N=68) | Placebo (N=65)
Injection site induration (General disorders) | 50 | 19
Injection site erythema (General disorders) | 31 | 11
Injection site pruritus (General disorders) | 20 | 9
Injection site pain (General disorders) | 18 | 2
Pyrexia (General disorders) | 10 | 4
Injection site swelling (General disorders) | 7 | 2
Malaise (General disorders) | 6 | 2
Oedema peripheral (General disorders) | 3 | 4
Nasopharyngitis (Infections and infestations) | 18 | 13
Upper respiratory tract infection (Infections and infestations) | 6 | 7
Herpes zoster (Infections and infestations) | 4 | 3
Pharyngitis (Infections and infestations) | 2 | 6
Bronchitis (Infections and infestations) | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 8 | 8
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 5
Stomatitis (Gastrointestinal disorders) | 2 | 7
Platelet count decreased (Investigations) | 7 | 9
Neutrophil count decreased (Investigations) | 1 | 5
Headache (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 3
Contusion (Injury, poisoning and procedural complications) | 2 | 4
Insomnia (Psychiatric disorders) | 2 | 4
Atrial fibrillation (Cardiac disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-07-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT01961882/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT01961882/SAP_001.pdf